CLINICAL TRIAL: NCT00549965
Title: A Multicenter, Prospective, Randomized, 2-Way Crossover, Open-Label Phase IV Study in Postmenopausal Women With Osteoporosis Examining Subject Satisfaction and Compliance When Actonel(Rosedronate) is Administered 35mg Once a Week or 5mg
Brief Title: Satisfaction and Compliance of Risedronate in PMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HMR4003B_4035
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-10

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

INTERVENTIONS:
Drug: Risedronate Sodium

SUMMARY:
Compare subject satisfaction of once a week dosing of 35 mg Risedronate to once daily dosing of 5 mg Risedronate in postmenopausal osteoporotic women. Secondary objectives are to measure compliance (50 % drug taken), and persistence.

ELIGIBILITY:
Inclusion Criteria:

* Five (5) years or greater postmenopausal who present with a diagnosis of postmenopausal osteoporosis based on standard clinical practice criteria.
* Subjects must discontinue bisphosphonates, calcitonin, fluoride, glucocorticoids (> than or = to 5 mg prednisone or equivalent per day) and hormone replacement therapy including estrogen-related compounds at least 6 months prior to randomization. During the study, these drugs are not permitted other than the study medication, Risedronate.
* Other concomitant medications should be kept to a minimum, but if the drugs are considered necessary for the subject's welfare and are unlikely to interfere with study medication they may be given at the discretion of the Investigator.

Exclusion Criteria:

* Had a history of cancer within the past 5 years. Relatively benign skin malignancies, such as basal cell carcinoma or squamous cell carcinoma, are not an exclusion if the subject has been in remission for at least 6 months prior to enrollment.
* Diagnosis of hypocalcemia, hyperparathyroidism, and hyperthyroidism.
* History of alcohol and/or drug abuse.
* Subjects will be excluded for active gastrointestinal disease that may interfere with absorption or with ability to swallow an oral medication.
* Subjects will also be excluded for serious concurrent illness that would interfere with their ability to participate in the trial.
* Excluded medications: bisphosphonates, calcitonin or fluoride or hormone replacement therapy within the last 6 months.
* Known hypersensitivity to bisphosphonates and/or excipients.
* Abnormal laboratory parameters, which are clinically relevant according to the Investigator (including renal insufficiency; creatinine clearance < 30 mL/min)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2003-10

PRIMARY OUTCOMES:
Measurement of subject satisfaction of once a week 35 mg Risedronate and once daily 5 mg Risedronate. | A subject-administered questionnaire at 12 and 24 weeks will assess satisfaction.

SECONDARY OUTCOMES:
The subjects' compliance and persistence on treatment. Compliance as defined by more than 50% of the drug taken (by tablet count) during each Risedronate treatment period. | Persistence at week 12 and 24 will be defined as continuing Risedronate treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Choe Seong Choon, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Daegu, South Korea